CLINICAL TRIAL: NCT03997097
Title: Phosphodiesterase-type 5 Inhibitors in Adult and Adolescent Patients With Univentricular Heart Disease: a Multi-center, Randomized, Double Blind Phase III Study
Brief Title: Efficacy of Phosphodiesterase-type 5 Inhibitors in Patients With Univentricular Congenital Heart Disease
Acronym: VU-INHIB
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: New sponsor
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7574
Record Dates: First submitted 2019-06-18; First posted 2019-06-25 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Single-ventricle; Pulmonary Hypertension; Univentricular Heart
Keywords: Congenital heart defect; single ventricle; Pulmonary hypertension; sildenafil; pulmonary vasodilator; Eexercise capacity
MeSH Terms: conditions — Univentricular Heart; Hypertension, Pulmonary; Heart Defects, Congenital | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sildenafil (Experimental): • Patients randomised in the group 1 will receive sildenafil in 3 oral doses of 20 mg per day (t.i.d.), as defined in the marketing authorization indicated for PAH in adolescent and adult patients, and for a period of 6 months.
  Interventions: Drug: Sildenafil
- placebo (Placebo Comparator): • Patients in the group 2 will receive a placebo (t.i.d.), for the same period of 6 months. To guarantee the double blind, capsules will be similar in size and colour and will be differentiated only by a vial number regarding to the randomization list
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Sildenafil — Patients randomised in the group 1 will receive sildenafil in 3 oral doses of 20 mg per day
  Other Names: sildenafil group
  Arms: sildenafil
Drug: Placebos — Patients randomised in the group placebo in 3 oral doses of per day
  Other Names: placebo group
  Arms: placebo

SUMMARY:
In univentricular hearts, selective lung vasodilators such as phosphodiesterase type 5 (PDE5) inhibitors would decrease pulmonary resistance and improve exercise tolerance. However, the level of evidence for the use of PDE5 inhibitors in patients with a single ventricle (SV) remains limited. the investigators present the SV-INHIBITION study rationale, design and methods.The SV-INHIBITION trial is a nationwide multicentre, randomised, double blind, placebo-controlled, phase III study, aiming to evaluate the efficacy of sildenafil on the ventilatory efficiency during exercise, in teenagers and adult patients (>15 y.o.) with a SV. Patients with pulmonary arterial hypertension (mean pulmonary arterial pressure (mPAP) > 15 mmHg and trans-pulmonary gradient > 5 mmHg) measured by cardiac catheterisation, will be eligible. The primary outcome is the variation of the VE/VCO2 slope, measured by a cardiopulmonary exercise test, between baseline and 6 months of treatment. A total of 50 patients are required to observe a decrease of 5 ± 5 points in the VE/VCO2 slope, with a power of 90% power and an alpha risk of 5%. The secondary outcomes are: clinical outcomes, 6 minute walk test, SV function, NT Pro BNP, VO2max, stroke volume, mPAP, trans-pulmonary gradient, SF36 quality of life score, safety and acceptability. This study aims to answer the question whether PDE5 inhibitors should be prescribed in patients with a SV. This trial has been built focusing on the 3 levels of research defined by the WHO: disability (exercise tolerance), deficit (SV function), and handicap (quality of life).

DETAILED DESCRIPTION:
50 Patients with a single ventricle (e.g. univentricular heart), as defined by the ACC-CHD classification, with a mean pulmonary arterial pressure (mPAP) > 15 mmHg and a trans-pulmonary gradient (TPG) > 5 mmHg, and aged 15 years old and above, will be prospectively recruited in the participating centres during their regular follow-up.

Patients wil be randomised into 2 groups:

* Patients randomised in the group 1 will receive sildenafil in 3 oral doses of 20 mg per day (t.i.d.), as defined in the marketing authorization indicated for PAH in adolescent and adult patients, and for a period of 6 months.
* Patients in the group 2 will receive a placebo (t.i.d.), for the same period of 6 months. To guarantee the double blind, capsules will be similar in size and colour and will be differentiated only by a vial number regarding to the randomization list. The clinical trials unit of the sponsor's pharmacy will centralize treatment allocation and supply to the participating centres. Drug management (reception, storage, delivery and traceability) will be ensured by the pharmacies of the participating centres.

After the 6 month-treatment period, patients will be followed for 3 months, and undergo at least 2 safety visits (1 and 3 months after intervention, and if necessary, any supplementary unscheduled visits). In accordance with the recommendations of the drug notice, the treatment will be suspended progressively over 1 week (20 mg b.i.d for 3 days, then 20 mg q.d. for 4 days, and then stopped) with a reinforcement of the surveillance. Patients will be able to contact an emergency number during this period and the investigator may decide to continue open treatment with sildenafil if clinically justified.

The study will be conducted in compliance with the Good Clinical Practices protocol and Declaration of Helsinki principles. It was approved by a drawn National Ethics Committee (CPP) and by the French National Agency of Medicine and Health Products Safety (ANSM). Informed consent will be obtained from all patients and their parents or legal guardians for minors.

ELIGIBILITY:
Inclusion Criteria:

1. 15 years of age and over.
2. Patient's weight over 20 kg
3. Patients with CHD with a single ventricular type defined by the classification of congenital heart diseases in Orphanet (53).
4. PAH defined by diagnostic catheterization with mean PAP > 15 mmHg and a trans-pulmonary gradient > 5 mmHg, performed as part of the usual follow-up. No definition of PAH in SV is available as a result of a particular physiology. Therefore, we chose the 15mmHg cut-off, which is used in clinical routine to allow or contra-indicate the Fontan procedure [50,51].
5. Appropriate written informed consent (adult patients, legal parents for teenagers), and formal assent (teenagers), should to be provided.
6. Beneficiary of a health insurance.

Exclusion Criteria:

1. Patient who is unable to perform a cardio-pulmonary exercise test.
2. Cardiac surgery planned during the trial.
3. Patient treated by any pulmonary arterial vasodilator drug, as defined in the 2015 PH guidelines (52), within 6 months before inclusion, regardless the duration and the type(s) (oral, intravenous, subcutaneous, inhaled) of administration.
4. Patient treated by Sildenafil or any other type of phosphodiesterase-type 5 inhibitor (such as tadalafil) within 6 months before inclusion, regardless the duration of administration.
5. Interventional cardiac catheterization planned during the trial (collateral occlusion, fenestration occlusion, stenting, angioplasty, ablation of rhythm disorder), other than during the screening.
6. Participation in another clinical trial or administration of an off-label drug in the 4 weeks preceding the screening.
7. Pregnancy, desire for pregnancy, absence of contraception during the study period.
8. Severe hepatic insufficiency (Child-Pugh C class).
9. Hypersensitivity to the active substance or to any of the excipients of the tablet:

   microcrystalline cellulose, calcium hydrogen phosphate anhydrous, croscarmellose sodium, stearate of magnesium, hypromellose, titanium dioxide (E171), monohydrate lactose, glycerol triacetate.
10. Combination with products called "nitric oxide donors" (such as amyl nitrite) or with nitrates in any form, due to the hypotensive effects of nitrates.
11. Concomitant administration of PDE5 inhibitors, such as Sildenafil, with guanylate cyclase stimulators, such as Riociguat.
12. Combination with the most potent inhibitors of CYP3A4 (eg ketoconazole, itraconazole, ritonavir).
13. Disposition to priapism, sclerosis of corpora cavernosa, disease of La Peyronie, sickle cell anemia, multiple myeloma, leukemia.
14. Uncontrolled hypotension or risk of hypotension: water depletion, obstruction to ejection of the left ventricle, dysfunction of the autonomic nervous system, patient under alpha-blocker.
15. Severe cardiovascular events, recent (<3 months) or not stabilized: myocardial infarction, unstable angina, sudden cardiac death, ventricular arrhythmia, cerebrovascular hemorrhage.
16. Active hemorrhagic disorders.
17. Active gastro-duodenal ulcer.
18. Patients with loss of vision of an eye due to non-arteritic anterior ischemic optic neuropathy (NAION), whether or not this event has been associated with previous exposure to a PDE5 inhibitor.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
ventilatory efficiency M0 | Month 0
  ventilatory efficiency, e.g. the VE/VCO2 slope, measured by CPET
ventilatory efficiency M6 | Month 6
  ventilatory efficiency, e.g. the VE/VCO2 slope, measured by

SECONDARY OUTCOMES:
VO2 max M0 | Month 0
  maximum oxygen uptake mesured by Cardio-pulmonary exercise test (CPET)
VO2 max M6 | Month 6
  maximum oxygen uptake mesured by Cardio-pulmonary exercise test (CPET)
ventilatory anaerobic threshold M0 | Month 0
  VAT using Beaver's method
ventilatory anaerobic threshold M6 | Month 6
  VAT using Beaver's method
oxygen pulse M0 | Month 0
  ratio VO2/heart rate M0
oxygen pulse M6 | Month 6
  ratio VO2/heart rate M6
OUES M0 | Month 0
  oxygen uptake efficiency slope mesured by CPET
OUES M6 | Month 6
  oxygen uptake efficiency slope mesured by CPET
NYHA functional class M0 | Month 0
  Functional class from I to IV (New York Heart Association Functional classification).
NYHA functional class M6 | Month 6
  Functional class from I to IV (New York Heart Association Functional classification).
blood pressure M0 | Month 0
  SV function evaluation with non-invasive imaging
blood pressure M6 | Month 6
  function evaluation with non-invasive imaging
oxygen saturation SaO2 | Month 0
  oxygen saturation measured using a transcutaneous sensor
oxygen saturation SaO2 | Month 6
  oxygen saturation measured using a transcutaneous sensor
6-minute walk test (6MWT) | Month 0
  6-minute walk test
6-minute walk test (6MWT) | Month 6
  6-minute walk test
Health-related quality of life | Month 0
  The SF-36 questionnaire
Health-related quality of life | Month 6
  The SF-36 questionnaire
Systemic blood flow | Month 0
  SV function with echocardiography
Systemic blood flow | Month 6
  SV function with echocardiography
SV systolic ejection fraction | Month 0
  SV function with echocardiography
SV systolic ejection fraction | Month 6
  SV function with echocardiography
2D strain SV function | Month 0
  SV function with echocardiography
2D strain SV function | Month 6
  SV function with echocardiography
Systemic blood flows in phase contrast | Month 0
  SV function evaluation with MRI
Systemic blood flows in phase contrast | Month 6
  SV function evaluation with MRI
Pulmonary blood flows in phase contrast | Month 0
  SV function evaluation with MRI
Pulmonary blood flows in phase contrast | Month 6
  SV function evaluation with MRI
SV systolic ejection fraction | Month 0
  SV function evaluation with MRI
SV systolic ejection fraction | Month 6
  SV function evaluation with MRI
SV systolic ejection volume | Month 0
  SV function evaluation with MRI
SV systolic ejection volume | Month 6
  SV function evaluation with MRI
NT Pro BNP | Month 0
  blood test checked
NT Pro BNP | Month 6
  blood test checked
forced expiratory volume in 1 s (FEV1 ) | month 0
  FEV1 spirometry
forced expiratory volume in 1 s (FEV1 ) | month 6
  FEV1 spirometry
Forced vital capacity FVC | month 0
  FVC spirometry
Forced vital capacity FVC | month 6
  FVC spirometry
FEV1% | month 0
  FEV1/FEVC ratio
FEV1% | month 6
  FEV1/FEVC ratio
DEMM25/75 | month 0
  DEMM25/75 measured by spirometry
DEMM25/75 | month 6
  DEMM25/75 measured by spirometry
Capillary lung volume | month 0
  pulmonary CO/NO transfer (patient seated and lying down)
Capillary lung volume | month 6
  pulmonary CO/NO transfer (patient seated and lying down)
Cardiac catheterization | month 0
  pulmonary arterial pressure mmHg
Cardiac catheterization | month 6
  pulmonary arterial pressure mmHg
percentage of patients compliant at 6 months of study treatment | month 6
  percentage of patients compliant
AE | month 6
  type of Averse events
SAE | month 6
  type of serious Averse events

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AMEDRO, MD, PhD, Principal Investigator — University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amedro P, Gavotto A, Abassi H, Picot MC, Matecki S, Malekzadeh-Milani S, Levy M, Ladouceur M, Ovaert C, Aldebert P, Thambo JB, Fraisse A, Humbert M, Cohen S, Baruteau AE, Karsenty C, Bonnet D, Hascoet S; SV-INHIBITION study investigators. Efficacy of phosphodiesterase type 5 inhibitors in univentricular congenital heart disease: the SV-INHIBITION study design. ESC Heart Fail. 2020 Apr;7(2):747-756. doi: 10.1002/ehf2.12630. Epub 2020 Mar 9. PMID 32147955